CLINICAL TRIAL: NCT04661813
Title: Assess and Adapt to the Impact of COVID-19 on CVD Self-Management and Prevention Care in Adults Living With HIV
Acronym: AAIM-High
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Duke University (Other); Metro Health, Michigan (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University Hospitals Cleveland Medical Center (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Chris Todd Longenecker, Associate Professor of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 03-18-16-S1; U01HL142099 (NIH)
Record Dates: First submitted 2020-10-29; First posted 2020-12-10 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: HIV-1-infection; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Single arm hybrid type 3 implementation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXTRA-CVD Virtual Care (Experimental): An adapted version of a "Nurse-led intervention to EXtend the HIV TReatment CascAde for CardioVascular Disease prevention" (EXTRA-CVD).
  Interventions: Other: EXTRA-CVD Virtual Care

INTERVENTIONS:
Other: EXTRA-CVD Virtual Care — The original EXTRA-CVD intervention was developed to improve blood pressure and cholesterol control among People Living with HIV. The intervention will be adapted to the post-COVID healthcare delivery landscape as a "virtual" intervention delivered by phone, teleconference, internet support groups, and nurse care coordination.

SUMMARY:
Social distancing measures put in place to combat the COVID-19 disease pandemic may increase social isolation and impact cardiovascular disease prevention behaviors among people living with HIV (PLWH). This study builds on a previously developed nurse-led intervention to improve blood pressure and cholesterol care for PLWH. The investigators will adapt the intervention to be administered virtually in order to facilitate cardiovascular prevention care within the US health care system which has sustained long-term changes as a result of the COVID-19 pandemic. The implementation and effectiveness of the intervention will be tested in a 12-month single arm intervention study.

DETAILED DESCRIPTION:
Social distancing in the context of the SARS-CoV-2 coronavirus and COVID-19 disease pandemic may amplify isolation and loneliness due to the requirement to limit in-person interactions with loved ones, friends, community members, healthcare providers, etc. Social isolation increases susceptibility to illness, stress, hypertension, depression, and mortality and decreases engagement in self-management and physical activity. People living with HIV (PLWH) are at increased risk for cardiovascular disease (CVD) and are particularly vulnerable to the stress and social isolation caused by the public health measures to combat COVID-19. Using mixed-methods and a human-centered design approach, the investigators will adapt a nurse-led intervention to EXtend the HIV/AIDS TReatment cAscade for CVD prevention (EXTRA-CVD) so that it is better suited to a post-COVID healthcare environment. This hybrid type 3 implementation study will evaluate the implementation of a virtually enhanced EXTRA-CVD intervention to improve BP control in PLWH from 3 HIV-specialty clinics in the United States [University Hospitals, MetroHealth (both Cleveland, OH) and Duke Health (Durham, NC)]. The study will enroll adult PLWH participants (n=75) on suppressive ART with high blood pressure whom are otherwise ineligible for the parent trial (EXTRA-CVD; NCT03643705) because they do not also have high cholesterol or because they are unwilling or unable to participate in the in-person trial. Primary outcomes will be: reach (% agreeing to participate), effectiveness (change in home systolic BP), and adoption (frequency of home BP use). Additional implementation measures including feasibility, acceptability, and intention to maintain blood pressure self-monitoring will be assessed qualitatively. This study will increase the impact and scalability of the EXTRA-CVD intervention without compromising the integrity or feasibility of the parent trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Confirmed HIV+ diagnosis
3. Undetectable HIV viral load: defined as the most recent HIV viral load <200 copies/mL, checked within the past year (assessed via chart abstraction)
4. Hypertension: defined as systolic BP >130 mmHg on ≥ 2 occasions in the past 12 months or on an antihypertensive medication (assessed via chart abstraction), and

Exclusion Criteria:

1. On anti-hypertensive medications solely for a non-hypertension indication (e.g. systolic heart failure),
2. Severely hearing or speech impaired, or other disability that would limit participation in the intervention components, and
3. In a nursing home and/or receiving in-patient psychiatric care.
4. Terminal illness with life expectancy < 4 months
5. No reliable access to a telephone
6. Pregnant, breast-feeding, or planning a pregnancy during the study period
7. Planning to move out of the area in the next 12 months
8. Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris T Longenecker, MD, Principal Investigator — University of Washington; Allison Webel, RN, PhD, Principal Investigator — University of Washington; Hayden Bosworth, PhD, Principal Investigator — Duke University; Barb Gripshover, MD, Principal Investigator — Case Western Reserve University
Locations (3):
- United States (3):
  - Duke Health, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
In collaboration with the National Institutes of Health funding body, we will develop a process to facilitate providing other investigators with access to appropriately de-identified study data. We will make the following available upon request after the primary manuscript is published: de-identified data set, trial description information, data collection forms, and data structure.
Time Frame: After publication of the primary manuscript
Access Criteria: Data will be made available upon request or on a data share site after publication of the primary manuscript.

REFERENCES:
- [Background] Okeke NL, Webel AR, Bosworth HB, Aifah A, Bloomfield GS, Choi EW, Gonzales S, Hale S, Hileman CO, Lopez-Kidwell V, Muiruri C, Oakes M, Schexnayder J, Smith V, Vedanthan R, Longenecker CT. Rationale and design of a nurse-led intervention to extend the HIV treatment cascade for cardiovascular disease prevention trial (EXTRA-CVD). Am Heart J. 2019 Oct;216:91-101. doi: 10.1016/j.ahj.2019.07.005. Epub 2019 Jul 18. PMID 31419622

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 81 participants consented to participate in the study. Of these, 7 participants withdrew prior to completion of the entry visit data collection, leaving 74 participants who actually started the study.
Period: Overall Study
Arm/Group | EXTRA-CVD Virtual Care
Started | 74 (This number differs from the 81 participants who consented because 7 participants withdrew prior to starting the study.)
Completed | 55
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | EXTRA-CVD Virtual Care
Number analyzed (Participants) | 74
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [51 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 45
  White | 24
  More than one race | 3
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 74
Enrollment site [Count of Participants; unit: Participants] — Site specific information is reported anonymously.
  Participants
    Site A | 24
    Site B | 25
    Site C | 25

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eligible Participants Who Agree to Participate
Description: Monitored continuously during study enrollment period
Time Frame: Through completion of study enrollment, an average of 9 months
Population: Total number of eligible patients based on telephone screen
Measure: Count of Participants; unit: Participants
Arm/Group | EXTRA-CVD Virtual Care
Number analyzed (Participants) | 103
Participants | 74

2. Primary Outcome: Average of Home Blood Pressure Values Assessed Over a 2-week Period at 0-, 4-, 8-, and 12-months.
Description: Repeated measures analysis across 4 time-points (0-, 4-, 8-, and 12-months)
Time Frame: 12 months
Population: Only participants who recorded blood pressure measurements at home during the 2-week period prior to their visit are included in the analysis. This explains why the number of participants analyzed is lower than the overall total number of study participants.
Measure: Mean (Standard Error); unit: model estimated mmhg
Groups:
- Baseline: Model-estimated mean home systolic BP over initial 2 week period of the study.
- 4 Months: Model-estimated mean home systolic BP through 4 months
- 8 Months: Model-estimated mean home systolic BP through 8 months
- 12 Months: Model-estimated mean home systolic BP through 12 months
Arm/Group | Baseline | 4 Months | 8 Months | 12 Months
Number analyzed (Participants) | 64 | 57 | 40 | 41
model estimated mmhg | 134.3 (1.5) | 128.9 (1.6) | 127.6 (1.8) | 126.5 (1.8)

3. Primary Outcome: Number of Days With at Least 1 Home Blood Pressure Measurement Assessed Over a 2-week Period at 0-, 4-, 8-, and 12-months.
Description: Repeated measures analysis across 4 time-points (0-, 4-, 8-, and 12-months)
Time Frame: 12 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Baseline: Number of days with at least one blood pressure measurement over the initial 2 week period
- 4 Months: Numbers of days with at least one home blood pressure measurement over a two week period preceding the 4 month visit
- 8 Months: Numbers of days with at least one home blood pressure measurement over a two week period preceding the 8 month visit
- 12 Months: Numbers of days with at least one home blood pressure measurement over a two week period preceding the 12 month visit
Arm/Group | Baseline | 4 Months | 8 Months | 12 Months
Number analyzed (Participants) | 64 | 57 | 40 | 41
days | 7 [4.5 to 10] | 7 [4 to 10] | 7.5 [5 to 12.5] | 7 [6 to 13]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events data were collected by study nurses through a combination of chart review and participant self report at baseline, 0-, 4-, 8-, and 12-months. The numbers reported here reflect the total number of AEs over the 12 month study period
Arm/Group | EXTRA-CVD Virtual Care
All-Cause Mortality (participants affected / at risk) | 3/74
Serious Adverse Events (participants affected / at risk) | 10/74
Other Adverse Events (participants affected / at risk) | 28/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EXTRA-CVD Virtual Care (N=74)
Non-study related events (General disorders) | 8 (16)
Hospitalization for bradycardia and syncope (Cardiac disorders) | 1 (1)
Emergency room visit for elevated home blood pressure (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EXTRA-CVD Virtual Care (N=74)
Non-study related events (General disorders) | 25 (40)
Asymptomatic hypotension (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1) — Fatigue, anorexia and malaise after starting lisinopril and hydrochlorothiazide
Lightheadedness (Cardiac disorders) | 1 (1) — Lightheadedness with new amlodipine dose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT04661813/Prot_SAP_001.pdf